CLINICAL TRIAL: NCT00223314
Title: HIV Prevention Among Alternative School Youth
Brief Title: Safer Choices 2 - HIV, STD, & Pregnancy Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Susan Tortolero/ Associate Professor and Director of the Center for Health Promotion & Prevention Research, University of Texas Houston School of Public Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HD038457-01 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: HIV; Sexually Transmitted Diseases; Pregnancy; HIV Infections
Keywords: HIV; Sexually Transmitted Diseases; Pregnancy; HIV Seronegativity
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections | interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: HIV, STD, Pregnancy Prevention Curriculum — The curriculum is designed to change students' knowledge, perceptions of norms, beliefs, self-efficacy, interpersonal skills (i.e., refusal skills), and high-risk behaviors related to HIV. The curriculum included use of facilitators for selected lessons such as role playing. Intervention strategies included demonstrations of skills by role playing, use of role model stories, and other experiential learning techniques. The curriculum was delivered during the school days by facilitators (project staff) who received intensive training prior to implementation and coaching and support during implementation.
  Other Names: Safer Choices 2

SUMMARY:
The purpose of the study is to adapt, implement, and evaluate an effective theoretically-based, high school HIV prevention program,Safer Choices, for higher risk youth in alternative schools.

Primary Research Question

1. Did the intervention reduce the number of occasions of unprotected sexual intercourse, number of sexual partners, and the proportion of students currently sexually active among those receiving the multiple component intervention relative to those students in the comparison group?

DETAILED DESCRIPTION:
This is a group-randomized intervention trial to reduce sexual risk-taking behaviors among young people attending alternative schools with a slight modification in the typical, group-randomized study design.

We will conduct the study in two waves. For Wave One, we will randomize 10 alternative schools (5 to intervention and 5 to comparison conditions), and then recruit and enroll a cohort of 500, 9th-grade students into the study (cohort 1). For Wave Two, we will cross-over the treatment conditions among the schools and enroll a new cohort of 9th-grade students into the study. Prior to the intervention, we will conduct a baseline measurement and conduct a post-intervention measurement at 6-, 12- and 24-months. The major hypothesis to be tested is that adolescents attending alternative schools who receive a multi-component HIV/STD intervention will reduce levels of unprotected sexual intercourse relative to those in the comparison condition. The major dependent variables are unprotected sexual intercourse, number of sexual partners, and proportion currently sexually active (last 3 months).

The specific aims of this project are to:

1. Adapt a tested, school-based, multi-component HIV prevention intervention for high-risk adolescents attending alternative schools using qualitative data from the target population and community representatives.
2. Assess the community acceptance, cultural sensitivity, and relevance of the proposed program for the target population.
3. Evaluate the effect of the multi-component HIV intervention on sexual risk-taking behaviors (unprotected sexual intercourse, number of sexual partners, deciding not to have sexual intercourse) among high-risk youth attending alternative schools.
4. Evaluate the effect of the multi-component HIV intervention on decreasing other risk-taking behaviors such as substance use and needle sharing behavior among youth attending alternative schools.
5. Evaluate the effect of the multi-component HIV intervention on student impact variables such as knowledge, self efficacy, attitudes, barriers, and perceived norms among youth attending alternative schools.
6. Disseminate findings to the scientific community, school districts, and community agencies.

We will conduct this study among 9th- grade students attending alternative schools in Houston Independent School District (HISD) and other community alternative schools. HISD Central Administration and Community Education Partners, the major HISD contractor, for alternative schools have agreed to participate in the study. We have identified ten alternative schools that have agreed to participate in the study. Students who are enrolled in alternative schools are fairly heterogeneous in terms of the rationale for being in these types of programs. Students may be in these programs for a variety of reasons including, low school performance, high absenteeism, truancy, behavior problems, social problems, pregnancy, or being in the juvenile justice system. However, all of the students enrolled in the identified schools are considered high-risk adolescents. We have identified 10 schools that have agreed to participate in the study with a total number of students enrolled in 9th grade at over 1000 students per year providing a more than adequate target population for recruitment. Of these students, 36% are African-American and 60% are Hispanic. Approximately 43% of the population are female.

Parental and student consent will be secured prior to administration of the risk assessment. Procedures will be used to achieve high rates of parental consent including sending information home about the project with particular emphasis on the confidential nature of the risk assessment.

Risk assessment data will be collected by using a talking, interactive computer for the collection of baseline, 6-month, 12-month, and 24-month post-intervention followup.

Baseline data collection will be conducted in the schools. The data collection staff will give a brief overview of how to use the computer and will help them to enter basic demographic information to acquaint them with the procedures. The computer will be equipped with headphones to maintain privacy, and the respondent can ask questions to our data collection staff, if needed. Post-intervention risk assessments will be conducted in the schools as youth are still enrolled in the alternative school program. We expect that the majority of students will still be enrolled in the alternative school at the 6-month followup, but that the 12-month and 24-month follow up will have to be conducted in various locations. We will track students enrolled in the study and conduct their follow up assessments in school, home, or in a location that is mutually agreed upon.

Curriculum Component We will adapt an existing curriculum, Safer Choices, to high-risk alternative school youth by obtaining feedback from the target population, conducting focus groups with parents and youths, and by obtaining feedback from community agencies through the Community Advisory Board. Although, Safer Choices was found to be effective in reducing unprotected sexual intercourse among inner-city high school students in Houston, the curriculum may need to be adapted to the experiences of these alternative school youth.

The target population has much higher prevalence of risk behaviors at younger ages than adolescents in regular schools.Further, these youth are at much greater risk of abusing drugs, being involved with legal authorities, being from single family households, having lower social support, having academic difficulties and learning disabilities, having suicide ideation and depression, and living in poorer communities. In adapting the program, therefore, we face the challenge of making the program fit the setting and students in alternative schools.

The curriculum will be designed to change students' knowledge, perceptions of norms, beliefs, self-efficacy, interpersonal skills (i.e., refusal skills), and high-risk behaviors related to HIV. The curriculum will include use of peer facilitators for selected lessons such as role playing. Intervention strategies will include demonstrations of skills by role playing, use of role model stories, and other experiential learning techniques. The Safer Choices curriculum will be modified to combine the 9th and 10th grade lessons to select those lessons which best match with the learning objectives for high-risk youth. The curriculum will be delivered during the school days by facilitators (project staff) who will receive intensive training prior to implementation and coaching and support during implementation. The Teacher Training Protocol used for Safer Choices will be adapted to train facilitators.

ELIGIBILITY:
Inclusion Criteria:

* 7th grade to 12 grade
* Attend one of the ten recruited schools

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2000-11; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Among those reporting intercourse: # of occasions students had unprotected sexual intercourse and # of sexual partners with whom students had unprotected intercourse; proportion of students initiating sexual intercourse in the past 3 months. | 24 months

SECONDARY OUTCOMES:
Alcohol use behavior: frequency of drinking alcohol or being drunk before having sexual intercourse in the past three months. | 24 months
Drug use behavior: frequency of other drug use before having sex in the past three months. | 24 moths
Drug use behavior: frequency of needle-sharing behavior during the past 12 months (one item). | 24 months
Number of lifetime tests for HIV infection, | 24 months
Number of lifetime tests for STD infection other than HIV. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Tortolero, PhD, Principal Investigator — University of TExas Houston Health Science Center-School of Public Health; Soledad L Escobar-Chaves, DrPH, Study Director — University of Texas Houston Health Science Center- School of Public Health
Locations (1):
- University of Texas Houston Health Science Center - School of Public Health, Houston, Texas, United States

REFERENCES:
- [Result] Escobar-Chaves SL, Tortolero SR, Markham C, Kelder SH, Kapadia A. Violent behavior among urban youth attending alternative schools. J Sch Health. 2002 Nov;72(9):357-62. doi: 10.1111/j.1746-1561.2002.tb03559.x. PMID 12557630
- [Result] Peters RJ Jr, Tortolero SR, Addy RC, Markham C, Escobar-Chaves SL, Fernandez-Esquer M, Yacoubian GS Jr. The relationship between sexual abuse and drug use: findings from Houston's Safer Choices 2 program. J Drug Educ. 2003;33(1):49-59. doi: 10.2190/3J7L-YN0E-JAJ8-QC6P. PMID 12773024
- [Result] Buzi RS, Tortolero SR, Roberts RE, Ross MW, Markham CM, Fleschler M. Gender differences in the consequences of a coercive sexual experience among adolescents attending alternative schools. J Sch Health. 2003 May;73(5):191-6. doi: 10.1111/j.1746-1561.2003.tb03602.x. PMID 12793105
- [Result] Peters RJ Jr, Tortolero SR, Addy RC, Markham C, Yacoubian GS Jr, Escobar-Chaves LS. Drug use among Texas alternative school students: findings from Houston's Safer Choices 2 Program. J Psychoactive Drugs. 2003 Jul-Sep;35(3):383-7. doi: 10.1080/02791072.2003.10400022. PMID 14621137
- [Result] Buzi RS, Tortolero SR, Roberts RE, Ross MW, Addy RC, Markham CM. The impact of a history of sexual abuse on high-risk sexual behaviors among females attending alternative schools. Adolescence. 2003 Winter;38(152):595-605. PMID 15053488
- [Result] Tortolero SR, Markham CM, Parcel GS, Peters RJ Jr, Escobar-Chaves SL, Basen-Engquist K, Lewis HL. Using intervention mapping to adapt an effective HIV, sexually transmitted disease, and pregnancy prevention program for high-risk minority youth. Health Promot Pract. 2005 Jul;6(3):286-98. doi: 10.1177/1524839904266472. PMID 16020623
- [Result] Markham CM, Tortolero SR, Escobar-Chaves SL, Parcel GS, Harrist R, Addy RC. Family connectedness and sexual risk-taking among urban youth attending alternative high schools. Perspect Sex Reprod Health. 2003 Jul-Aug;35(4):174-9. doi: 10.1363/psrh.35.174.03. PMID 12941650